CLINICAL TRIAL: NCT00089791
Title: A Study to Evaluate Denosumab in the Treatment of Postmenopausal Osteoporosis FREEDOM (Fracture REduction Evaluation of Denosumab in Osteoporosis Every 6 Months)
Brief Title: A Study to Evaluate Denosumab in the Treatment of Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20030216
Record Dates: First submitted 2004-08-13; First posted 2004-08-16 (Estimated); Results first posted 2014-01-10 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Osteoporosis
Keywords: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo administered subcutaneously once every 6 months for 3 years.
  Interventions: Drug: placebo
- Denosumab 60 mg Q6M (Experimental): Denosumab 60 mg administered subcutaneously once every 6 months (Q6M) for 3 years.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: placebo — Placebo administered by subcutaneous injection
  Arms: Placebo
Drug: Denosumab — Denosumab 60 mg administered by subcutaneous injection
  Other Names: AMG 162; Prolia®
  Arms: Denosumab 60 mg Q6M

SUMMARY:
This study will evaluate the effectiveness and safety of denosumab in treating women with Postmenopausal Osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 60 to 90 years of age may be eligible to participate
* Bone mineral density (BMD) T-Score at hip or spine must be less than -2.5

Exclusion Criteria:

* BMD T-Score at the hip or the spine of less than -4.0
* Patients with any severe or more than two moderate vertebral fractures on spinal x-ray at entry

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7808 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2008-06-17 (Actual); Study Completion 2008-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Adami S, Libanati C, Boonen S, Cummings SR, Ho PR, Wang A, Siris E, Lane J; FREEDOM Fracture-Healing Writing Group; Adachi JD, Bhandari M, de Gregorio L, Gilchrist N, Lyritis G, Moller G, Palacios S, Pavelka K, Heinrich R, Roux C, Uebelhart D. Denosumab treatment in postmenopausal women with osteoporosis does not interfere with fracture-healing: results from the FREEDOM trial. J Bone Joint Surg Am. 2012 Dec 5;94(23):2113-9. doi: 10.2106/JBJS.K.00774. PMID 23097066
- [Background] Austin M, Yang YC, Vittinghoff E, Adami S, Boonen S, Bauer DC, Bianchi G, Bolognese MA, Christiansen C, Eastell R, Grauer A, Hawkins F, Kendler DL, Oliveri B, McClung MR, Reid IR, Siris ES, Zanchetta J, Zerbini CA, Libanati C, Cummings SR; FREEDOM Trial. Relationship between bone mineral density changes with denosumab treatment and risk reduction for vertebral and nonvertebral fractures. J Bone Miner Res. 2012 Mar;27(3):687-93. doi: 10.1002/jbmr.1472. PMID 22095631
- [Background] Bolognese MA, Teglbjaerg CS, Zanchetta JR, Lippuner K, McClung MR, Brandi ML, Hoiseth A, Lakatos P, Moffett AH, Lorenc RS, Wang A, Libanati C. Denosumab significantly increases DXA BMD at both trabecular and cortical sites: results from the FREEDOM study. J Clin Densitom. 2013 Apr-Jun;16(2):147-53. doi: 10.1016/j.jocd.2012.02.006. Epub 2012 Apr 20. PMID 22521543
- [Background] Boonen S, Adachi JD, Man Z, Cummings SR, Lippuner K, Torring O, Gallagher JC, Farrerons J, Wang A, Franchimont N, San Martin J, Grauer A, McClung M. Treatment with denosumab reduces the incidence of new vertebral and hip fractures in postmenopausal women at high risk. J Clin Endocrinol Metab. 2011 Jun;96(6):1727-36. doi: 10.1210/jc.2010-2784. Epub 2011 Mar 16. PMID 21411557
- [Background] Brown JP, Roux C, Torring O, Ho PR, Beck Jensen JE, Gilchrist N, Recknor C, Austin M, Wang A, Grauer A, Wagman RB. Discontinuation of denosumab and associated fracture incidence: analysis from the Fracture Reduction Evaluation of Denosumab in Osteoporosis Every 6 Months (FREEDOM) trial. J Bone Miner Res. 2013 Apr;28(4):746-52. doi: 10.1002/jbmr.1808. PMID 23109251
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Background] Eastell R, Christiansen C, Grauer A, Kutilek S, Libanati C, McClung MR, Reid IR, Resch H, Siris E, Uebelhart D, Wang A, Weryha G, Cummings SR. Effects of denosumab on bone turnover markers in postmenopausal osteoporosis. J Bone Miner Res. 2011 Mar;26(3):530-7. doi: 10.1002/jbmr.251. PMID 20839290
- [Background] Freemantle N, Cooper C, Diez-Perez A, Gitlin M, Radcliffe H, Shepherd S, Roux C. Results of indirect and mixed treatment comparison of fracture efficacy for osteoporosis treatments: a meta-analysis. Osteoporos Int. 2013 Jan;24(1):209-17. doi: 10.1007/s00198-012-2068-9. Epub 2012 Jul 26. PMID 22832638
- [Background] Genant HK, Libanati C, Engelke K, Zanchetta JR, Hoiseth A, Yuen CK, Stonkus S, Bolognese MA, Franek E, Fuerst T, Radcliffe HS, McClung MR. Improvements in hip trabecular, subcortical, and cortical density and mass in postmenopausal women with osteoporosis treated with denosumab. Bone. 2013 Oct;56(2):482-8. doi: 10.1016/j.bone.2013.07.011. Epub 2013 Jul 17. PMID 23871852
- [Background] Hadji P, Bock O, Resch H, Kraenzlin M, Wang A, Steinle T, Eisen C. Reduction of fracture risk with denosumab among women with osteoporosis with or without need for treatment according to DVO 2009 guideline : A subgroup analysis of the FREEDOM trial. Osteologie. 2013;22(1):39-45.
- [Background] Jamal SA, Ljunggren O, Stehman-Breen C, Cummings SR, McClung MR, Goemaere S, Ebeling PR, Franek E, Yang YC, Egbuna OI, Boonen S, Miller PD. Effects of denosumab on fracture and bone mineral density by level of kidney function. J Bone Miner Res. 2011 Aug;26(8):1829-35. doi: 10.1002/jbmr.403. PMID 21491487
- [Background] Keaveny TM, McClung MR, Genant HK, Zanchetta JR, Kendler D, Brown JP, Goemaere S, Recknor C, Brandi ML, Eastell R, Kopperdahl DL, Engelke K, Fuerst T, Radcliffe HS, Libanati C. Femoral and vertebral strength improvements in postmenopausal women with osteoporosis treated with denosumab. J Bone Miner Res. 2014 Jan;29(1):158-65. doi: 10.1002/jbmr.2024. PMID 23794225
- [Background] Mackey DC, Black DM, Bauer DC, McCloskey EV, Eastell R, Mesenbrink P, Thompson JR, Cummings SR. Effects of antiresorptive treatment on nonvertebral fracture outcomes. J Bone Miner Res. 2011 Oct;26(10):2411-8. doi: 10.1002/jbmr.446. PMID 21710615
- [Background] McCloskey EV, Johansson H, Oden A, Austin M, Siris E, Wang A, Lewiecki EM, Lorenc R, Libanati C, Kanis JA. Denosumab reduces the risk of osteoporotic fractures in postmenopausal women, particularly in those with moderate to high fracture risk as assessed with FRAX. J Bone Miner Res. 2012 Jul;27(7):1480-6. doi: 10.1002/jbmr.1606. PMID 22431426
- [Background] McClung MR, Boonen S, Torring O, Roux C, Rizzoli R, Bone HG, Benhamou CL, Lems WF, Minisola S, Halse J, Hoeck HC, Eastell R, Wang A, Siddhanti S, Cummings SR. Effect of denosumab treatment on the risk of fractures in subgroups of women with postmenopausal osteoporosis. J Bone Miner Res. 2012 Jan;27(1):211-8. doi: 10.1002/jbmr.536. PMID 21976367
- [Background] McClung MR, Zanchetta JR, Hoiseth A, Kendler DL, Yuen CK, Brown JP, Stonkus S, Goemaere S, Recknor C, Woodson GC, Bolognese MA, Franek E, Brandi ML, Wang A, Libanati C. Denosumab densitometric changes assessed by quantitative computed tomography at the spine and hip in postmenopausal women with osteoporosis. J Clin Densitom. 2013 Apr-Jun;16(2):250-6. doi: 10.1016/j.jocd.2012.02.014. Epub 2012 May 8. PMID 22572531
- [Background] Samelson EJ, Miller PD, Christiansen C, Daizadeh NS, Grazette L, Anthony MS, Egbuna O, Wang A, Siddhanti SR, Cheung AM, Franchimont N, Kiel DP. RANKL inhibition with denosumab does not influence 3-year progression of aortic calcification or incidence of adverse cardiovascular events in postmenopausal women with osteoporosis and high cardiovascular risk. J Bone Miner Res. 2014 Feb;29(2):450-7. doi: 10.1002/jbmr.2043. PMID 23873632
- [Background] Silverman S, Viswanathan HN, Yang YC, Wang A, Boonen S, Ragi-Eis S, Fardellone P, Gilchrist N, Lips P, Nevitt M, Palacios Gil-Antunano S, Pavelka K, Revicki D, Simon J, Macarios D, Siris ES. Impact of clinical fractures on health-related quality of life is dependent on time of assessment since fracture: results from the FREEDOM trial. Osteoporos Int. 2012 Apr;23(4):1361-9. doi: 10.1007/s00198-011-1720-0. Epub 2011 Jul 19. PMID 21769664
- [Background] Simon JA, Recknor C, Moffett AH Jr, Adachi JD, Franek E, Lewiecki EM, McClung MR, Mautalen CA, Ragi-Eis S, Nicholson GC, Muschitz C, Nuti R, Torring O, Wang A, Libanati C. Impact of denosumab on the peripheral skeleton of postmenopausal women with osteoporosis: bone density, mass, and strength of the radius, and wrist fracture. Menopause. 2013 Feb;20(2):130-7. doi: 10.1097/gme.0b013e318267f909. PMID 23010883
- [Background] Strom O, Jonsson B, Kanis JA. Intervention thresholds for denosumab in the UK using a FRAX(R)-based cost-effectiveness analysis. Osteoporos Int. 2013 Apr;24(4):1491-502. doi: 10.1007/s00198-012-2115-6. Epub 2012 Dec 7. PMID 23224141
- [Background] Watts NB, Roux C, Modlin JF, Brown JP, Daniels A, Jackson S, Smith S, Zack DJ, Zhou L, Grauer A, Ferrari S. Infections in postmenopausal women with osteoporosis treated with denosumab or placebo: coincidence or causal association? Osteoporos Int. 2012 Jan;23(1):327-37. doi: 10.1007/s00198-011-1755-2. Epub 2011 Sep 3. PMID 21892677
- [Derived] Hara T, Hijikata Y, Matsubara Y, Watanabe N. Pharmacological interventions versus placebo, no treatment or usual care for osteoporosis in people with chronic kidney disease stages 3-5D. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013424. doi: 10.1002/14651858.CD013424.pub2. PMID 34231877
- [Derived] Broadwell A, Chines A, Ebeling PR, Franek E, Huang S, Smith S, Kendler D, Messina O, Miller PD. Denosumab Safety and Efficacy Among Participants in the FREEDOM Extension Study With Mild to Moderate Chronic Kidney Disease. J Clin Endocrinol Metab. 2021 Jan 23;106(2):397-409. doi: 10.1210/clinem/dgaa851. PMID 33211870
- [Derived] Ferrari S, Lewiecki EM, Butler PW, Kendler DL, Napoli N, Huang S, Crittenden DB, Pannacciulli N, Siris E, Binkley N. Favorable skeletal benefit/risk of long-term denosumab therapy: A virtual-twin analysis of fractures prevented relative to skeletal safety events observed. Bone. 2020 May;134:115287. doi: 10.1016/j.bone.2020.115287. Epub 2020 Feb 21. PMID 32092479
- [Derived] Ferrari S, Eastell R, Napoli N, Schwartz A, Hofbauer LC, Chines A, Wang A, Pannacciulli N, Cummings SR. Denosumab in postmenopausal women with osteoporosis and diabetes: Subgroup analysis of FREEDOM and FREEDOM extension. Bone. 2020 May;134:115268. doi: 10.1016/j.bone.2020.115268. Epub 2020 Feb 10. PMID 32058020
- [Derived] Ferrari S, Butler PW, Kendler DL, Miller PD, Roux C, Wang AT, Huang S, Wagman RB, Lewiecki EM. Further Nonvertebral Fracture Reduction Beyond 3 Years for Up to 10 Years of Denosumab Treatment. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3450-3461. doi: 10.1210/jc.2019-00271. PMID 31125092
- [Derived] Watts NB, Grbic JT, Binkley N, Papapoulos S, Butler PW, Yin X, Tierney A, Wagman RB, McClung M. Invasive Oral Procedures and Events in Postmenopausal Women With Osteoporosis Treated With Denosumab for Up to 10 Years. J Clin Endocrinol Metab. 2019 Jun 1;104(6):2443-2452. doi: 10.1210/jc.2018-01965. PMID 30759221
- [Derived] Dempster DW, Brown JP, Fahrleitner-Pammer A, Kendler D, Rizzo S, Valter I, Wagman RB, Yin X, Yue SV, Boivin G. Effects of Long-Term Denosumab on Bone Histomorphometry and Mineralization in Women With Postmenopausal Osteoporosis. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2498-2509. doi: 10.1210/jc.2017-02669. PMID 29672714
- [Derived] Napoli N, Pannacciulli N, Vittinghoff E, Crittenden D, Yun J, Wang A, Wagman R, Schwartz AV. Effect of denosumab on fasting glucose in women with diabetes or prediabetes from the FREEDOM trial. Diabetes Metab Res Rev. 2018 May;34(4):e2991. doi: 10.1002/dmrr.2991. Epub 2018 Apr 16. PMID 29430796
- [Derived] Cummings SR, Ferrari S, Eastell R, Gilchrist N, Jensen JB, McClung M, Roux C, Torring O, Valter I, Wang AT, Brown JP. Vertebral Fractures After Discontinuation of Denosumab: A Post Hoc Analysis of the Randomized Placebo-Controlled FREEDOM Trial and Its Extension. J Bone Miner Res. 2018 Feb;33(2):190-198. doi: 10.1002/jbmr.3337. Epub 2017 Nov 22. PMID 29105841
- [Derived] Bone HG, Wagman RB, Brandi ML, Brown JP, Chapurlat R, Cummings SR, Czerwinski E, Fahrleitner-Pammer A, Kendler DL, Lippuner K, Reginster JY, Roux C, Malouf J, Bradley MN, Daizadeh NS, Wang A, Dakin P, Pannacciulli N, Dempster DW, Papapoulos S. 10 years of denosumab treatment in postmenopausal women with osteoporosis: results from the phase 3 randomised FREEDOM trial and open-label extension. Lancet Diabetes Endocrinol. 2017 Jul;5(7):513-523. doi: 10.1016/S2213-8587(17)30138-9. Epub 2017 May 22. PMID 28546097
- [Derived] Zebaze R, Libanati C, McClung MR, Zanchetta JR, Kendler DL, Hoiseth A, Wang A, Ghasem-Zadeh A, Seeman E. Denosumab Reduces Cortical Porosity of the Proximal Femoral Shaft in Postmenopausal Women With Osteoporosis. J Bone Miner Res. 2016 Oct;31(10):1827-1834. doi: 10.1002/jbmr.2855. Epub 2016 May 19. PMID 27082709
- [Derived] Reid IR, Miller PD, Brown JP, Kendler DL, Fahrleitner-Pammer A, Valter I, Maasalu K, Bolognese MA, Woodson G, Bone H, Ding B, Wagman RB, San Martin J, Ominsky MS, Dempster DW; Denosumab Phase 3 Bone Histology Study Group. Effects of denosumab on bone histomorphometry: the FREEDOM and STAND studies. J Bone Miner Res. 2010 Oct;25(10):2256-65. doi: 10.1002/jbmr.149. PMID 20533525
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 03-Aug-2004 Last Subject Enrolled: 01-Jun-2005
Period: Overall Study
Arm/Group | Placebo | Denosumab 60 mg Q6M
Started | 3906 | 3902
Received Study Medication | 3883 | 3879
Safety Analysis Set | 3876 (7 participants in the placebo arm received ≥1 dose of denosumab & were analyzed in the denosumab arm) | 3886
Completed | 3206 | 3272
Not Completed | 700 | 630
Not completed — Physician Decision | 6 | 3
Not completed — Adverse Event | 81 | 93
Not completed — Withdrawal by Subject | 403 | 344
Not completed — Death | 78 | 62
Not completed — Disease progression | 7 | 3
Not completed — Ineligibility determined | 12 | 9
Not completed — Lost to Follow-up | 57 | 57
Not completed — Noncompliance | 17 | 13
Not completed — Other | 20 | 32
Not completed — Protocol deviation | 12 | 10
Not completed — Requirement for alternative therapy | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Denosumab 60 mg Q6M | Total
Number analyzed (Participants) | 3906 | 3902 | 7808
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.3 (5.2) | 72.3 (5.2) | 72.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3906 | 3902 | 7808
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 3629 | 3609 | 7238
  Black or African American | 27 | 30 | 57
  Hispanic or Latino | 232 | 241 | 473
  Asian | 8 | 9 | 17
  Japanese | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Other | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New Vertebral Fractures
Description: A new vertebral fracture, assessed by lateral spine X-ray using Genant semiquantitative scoring method, was identified as an ≥ 1 grade increase from the Baseline grade of 0 in any vertebra from T4 to L4. New vertebral fractures included morphometric vertebral fractures (assessed at scheduled visits and not associated with signs or symptoms [or both] indicative of a fracture) and clinical vertebral fractures (assessed at either a scheduled or unscheduled visit and associated with any signs and/or symptoms indicative of a fracture, excluding any fracture associated with high trauma severity or a pathologic fracture).
Time Frame: 36 months
Population: Primary Efficacy Analysis Set, which includes all randomized participants who have a baseline and ≥ 1 postbaseline evaluation of vertebral fracture at or before 3 years. Last Observation Carried Forward was used.
Measure: Number; unit: Participants
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 3691 | 3702
Participants | 264 | 86
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, Mantel Haenszel — Logistic regression was used to generate the p-value; Risk Ratio (RR) = 0.32, 95% CI [0.26 to 0.41]

2. Secondary Outcome: Number of Participants With Nonvertebral Fractures
Description: Nonvertebral fractures (osteoporotic) were those occurring on study excluding those of the vertebrae (cervical, thoracic, and lumbar), skull, facial, mandible, metacarpus, finger phalanges, and toe phalanges. Fractures associated with high trauma severity (fractures that were the result of a fall from higher than the height of a stool, chair, first rung on a ladder or equivalent (> 20 inches) or was the result of severe trauma other than a fall) and pathologic fractures were excluded from this category. Nonvertebral fractures were required to be confirmed either by radiographs or other diagnostic images such as computerized tomography (CT) or magnetic resonance imaging (MRI), or by documentation in a radiology report, surgical report, or discharge summary.
Time Frame: 36 months
Population: Full analysis set (all randomized participants)
Measure: Number; unit: Participants
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 3906 | 3902
Participants | 293 | 238
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.0106, Regression, Cox; Hazard Ratio (HR) = 0.8, 95% CI [0.67 to 0.95]

3. Secondary Outcome: Number of Participants With a Hip Fracture
Description: Hip fractures are a subset of nonvertebral fractures including femur neck, femur intertrochanter, and femur subtrochanter.
Time Frame: 36 months
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Placebo | Denosumab 60 mg Q6M
Number analyzed (Participants) | 3906 | 3902
Participants | 43 | 26
Statistical Analysis 1: Comparison: Placebo vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p = 0.0362, Regression, Cox; Hazard Ratio (HR) = 0.6, 95% CI [0.37 to 0.97]

ADVERSE EVENTS:
Time Frame: 36 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events. Seven participants who were randomized to placebo but received denosumab in error are summarized in the denosumab arm.
Arm/Group | Placebo | Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 972/3876 | 1004/3886
Other Adverse Events (participants affected / at risk) | 3107/3876 | 3073/3886
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3876) | Denosumab 60 mg Q6M (N=3886)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 10 | 11
Anaemia megaloblastic (Blood and lymphatic system disorders) | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 1
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 6 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 3
Acute myocardial infarction (Cardiac disorders) | 5 | 12
Angina pectoris (Cardiac disorders) | 18 | 33
Angina unstable (Cardiac disorders) | 12 | 11
Aortic valve disease (Cardiac disorders) | 0 | 1
Aortic valve disease mixed (Cardiac disorders) | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 4
Arrhythmia (Cardiac disorders) | 5 | 4
Arteriosclerosis coronary artery (Cardiac disorders) | 3 | 4
Atrial fibrillation (Cardiac disorders) | 33 | 36
Atrial flutter (Cardiac disorders) | 3 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 3 | 3
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 3 | 4
Bundle branch block left (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 5 | 6
Cardiac failure (Cardiac disorders) | 15 | 16
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 5 | 1
Cardiac failure congestive (Cardiac disorders) | 13 | 10
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 4 | 1
Cardiogenic shock (Cardiac disorders) | 2 | 5
Cardiomegaly (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 17 | 15
Coronary artery insufficiency (Cardiac disorders) | 0 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 4
Coronary artery thrombosis (Cardiac disorders) | 0 | 3
Heart valve calcification (Cardiac disorders) | 1 | 0
Heart valve incompetence (Cardiac disorders) | 1 | 0
Hypertensive cardiomyopathy (Cardiac disorders) | 0 | 3
Hypertensive heart disease (Cardiac disorders) | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 2
Left ventricular failure (Cardiac disorders) | 3 | 2
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 23 | 25
Myocardial ischaemia (Cardiac disorders) | 5 | 12
Palpitations (Cardiac disorders) | 1 | 4
Pericardial haemorrhage (Cardiac disorders) | 0 | 2
Sick sinus syndrome (Cardiac disorders) | 4 | 9
Sinus arrhythmia (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 3 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 7
Tachyarrhythmia (Cardiac disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Tachycardia paroxysmal (Cardiac disorders) | 1 | 1
Ventricle rupture (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 2
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 2
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 | 1
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 1
Inner ear disorder (Ear and labyrinth disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 10 | 16
Vertigo positional (Ear and labyrinth disorders) | 1 | 1
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Vestibular neuronitis (Ear and labyrinth disorders) | 1 | 1
Goitre (Endocrine disorders) | 3 | 4
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 0
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Angle closure glaucoma (Eye disorders) | 0 | 2
Cataract (Eye disorders) | 28 | 21
Choroidal haemorrhage (Eye disorders) | 0 | 1
Corneal decompensation (Eye disorders) | 1 | 0
Dacryostenosis acquired (Eye disorders) | 2 | 1
Entropion (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 5
Keratitis (Eye disorders) | 0 | 1
Lens dislocation (Eye disorders) | 1 | 0
Macular degeneration (Eye disorders) | 5 | 3
Macular hole (Eye disorders) | 2 | 0
Myopia (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 3 | 3
Retinal disorder (Eye disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Retinal tear (Eye disorders) | 0 | 1
Retinal vascular thrombosis (Eye disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 2 | 1
Visual disturbance (Eye disorders) | 0 | 2
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 2 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 | 2
Acute abdomen (Gastrointestinal disorders) | 1 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anal polyp (Gastrointestinal disorders) | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Appendicitis perforated (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 4
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 3 | 1
Colonic haematoma (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 2
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 8 | 6
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 3 | 7
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 8
Duodenal ulcer (Gastrointestinal disorders) | 1 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocele (Gastrointestinal disorders) | 1 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 3 | 5
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 6 | 9
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 6
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 4
Hiatus hernia (Gastrointestinal disorders) | 3 | 4
Ileus (Gastrointestinal disorders) | 3 | 4
Inguinal hernia (Gastrointestinal disorders) | 5 | 7
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 2 | 2
Intestinal cyst (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 6
Intestinal perforation (Gastrointestinal disorders) | 1 | 1
Intussusception (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 3
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 2 | 1
Mesenteric artery embolism (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 5
Oesophagitis (Gastrointestinal disorders) | 0 | 3
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0
Pancreatic fistula (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 0 | 5
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Peritoneal haematoma (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 4
Pharyngoesophageal diverticulum (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 5
Rectal prolapse (Gastrointestinal disorders) | 2 | 6
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary gland cyst (Gastrointestinal disorders) | 0 | 1
Sigmoiditis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 2 | 1
Umbilical hernia (Gastrointestinal disorders) | 2 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 6
Accidental death (General disorders) | 2 | 1
Asthenia (General disorders) | 0 | 4
Cardiac death (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 3 | 3
Chills (General disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Death (General disorders) | 2 | 2
Fatigue (General disorders) | 1 | 1
Feeling hot (General disorders) | 1 | 1
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 1
Generalised oedema (General disorders) | 1 | 0
Hernia obstructive (General disorders) | 1 | 1
Impaired healing (General disorders) | 1 | 1
Inflammation (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 9 | 10
Oedema peripheral (General disorders) | 0 | 3
Pain (General disorders) | 2 | 1
Pelvic mass (General disorders) | 0 | 1
Polyp (General disorders) | 1 | 0
Pseudocyst (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 4
Sensation of pressure (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Ulcer haemorrhage (General disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 2 | 0
Biliary colic (Hepatobiliary disorders) | 2 | 0
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 3 | 4
Cholecystitis acute (Hepatobiliary disorders) | 4 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 17 | 17
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Chronic hepatitis (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Post cholecystectomy syndrome (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 2
Abscess intestinal (Infections and infestations) | 1 | 0
Acrodermatitis chronica atrophicans (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Appendiceal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 7 | 7
Arthritis viral (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Biliary tract infection fungal (Infections and infestations) | 0 | 1
Borrelia infection (Infections and infestations) | 0 | 1
Bronchiectasis (Infections and infestations) | 2 | 4
Bronchitis (Infections and infestations) | 7 | 4
Bronchopneumonia (Infections and infestations) | 7 | 6
Cellulitis (Infections and infestations) | 1 | 6
Cervicitis (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 2 | 1
Chronic sinusitis (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 1
Cystitis (Infections and infestations) | 2 | 6
Diverticulitis (Infections and infestations) | 6 | 8
Encephalitis viral (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 7
Escherichia infection (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastric infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 7 | 9
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1
Gastroenteritis bacterial (Infections and infestations) | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 2
Herpes zoster (Infections and infestations) | 2 | 1
Herpes zoster ophthalmic (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 4
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 2 | 0
Localised infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 6
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 2
Lung infection pseudomonal (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 1 | 0
Lymphangitis (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Phlebitis infective (Infections and infestations) | 0 | 1
Pleural infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 36 | 34
Pneumonia bacterial (Infections and infestations) | 2 | 2
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 3
Post procedural pneumonia (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 2 | 1
Pyelonephritis (Infections and infestations) | 2 | 5
Pyelonephritis acute (Infections and infestations) | 1 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Pyometra (Infections and infestations) | 0 | 1
Pyothorax (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 3
Respiratory tract infection fungal (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 4 | 3
Septic shock (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 3
Skin bacterial infection (Infections and infestations) | 0 | 2
Staphylococcal infection (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 1
Tubo-ovarian abscess (Infections and infestations) | 0 | 1
Typhus (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 10 | 16
Urosepsis (Infections and infestations) | 2 | 1
Vaginal infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic ulcer haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1 | 0
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Chemical eye injury (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 11 | 1
Contusion (Injury, poisoning and procedural complications) | 7 | 6
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 0 | 1
Device malfunction (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 1
Failure of implant (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 18 | 16
Femoral neck fracture (Injury, poisoning and procedural complications) | 20 | 13
Femur fracture (Injury, poisoning and procedural complications) | 28 | 14
Fibula fracture (Injury, poisoning and procedural complications) | 10 | 7
Foot fracture (Injury, poisoning and procedural complications) | 3 | 4
Fractured ischium (Injury, poisoning and procedural complications) | 1 | 2
Fractured sacrum (Injury, poisoning and procedural complications) | 2 | 1
Hand fracture (Injury, poisoning and procedural complications) | 2 | 1
Head injury (Injury, poisoning and procedural complications) | 9 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 13 | 11
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 6
Joint sprain (Injury, poisoning and procedural complications) | 1 | 2
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 9 | 3
Medical device complication (Injury, poisoning and procedural complications) | 4 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 7 | 4
Multiple injuries (Injury, poisoning and procedural complications) | 2 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 2 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 6 | 4
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Postoperative constipation (Injury, poisoning and procedural complications) | 0 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1
Radius fracture (Injury, poisoning and procedural complications) | 23 | 25
Retinal injury (Injury, poisoning and procedural complications) | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 5 | 6
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 2
Sciatic nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 3
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 9 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 10 | 6
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 17 | 7
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 1
Body temperature increased (Investigations) | 0 | 1
Cardiac murmur (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 1 | 0
Hepatic enzyme (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Intraocular pressure increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 1
Weight decreased (Investigations) | 4 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 7 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 5
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 3 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 20
Bone callus excessive (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Bunion (Musculoskeletal and connective tissue disorders) | 2 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondromalacia (Musculoskeletal and connective tissue disorders) | 1 | 0
Collagen disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 4 | 2
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 3 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 | 15
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Morphoea (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 79 | 63
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 3
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 3
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 5 | 6
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 | 5
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 10
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 3
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 2
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acral lentiginous melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 | 34
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Carcinoid tumour of the stomach (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 11
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 7
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 9
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymph node cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant lymphoid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to fallopian tube (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to large intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pseudolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Rectal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Schloffer tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urethral cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 2
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Brain stem ischaemia (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 5 | 1
Cauda equina syndrome (Nervous system disorders) | 0 | 2
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 2 | 2
Cerebral artery embolism (Nervous system disorders) | 1 | 1
Cerebral artery stenosis (Nervous system disorders) | 0 | 1
Cerebral circulatory failure (Nervous system disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 4 | 2
Cerebral infarction (Nervous system disorders) | 4 | 3
Cerebral ischaemia (Nervous system disorders) | 1 | 5
Cerebral thrombosis (Nervous system disorders) | 3 | 3
Cerebrovascular accident (Nervous system disorders) | 23 | 32
Cerebrovascular disorder (Nervous system disorders) | 2 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 2 | 1
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Cervicogenic headache (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 3 | 2
Dementia Alzheimer's type (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 7 | 5
Drop attacks (Nervous system disorders) | 1 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 3 | 2
Essential tremor (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 0 | 1
Global amnesia (Nervous system disorders) | 1 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 3
Hemianopia (Nervous system disorders) | 0 | 1
Hemicephalalgia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 8 | 7
Lacunar infarction (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 4 | 6
Lumbar radiculopathy (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 1 | 0
Miller Fisher syndrome (Nervous system disorders) | 0 | 1
Mononeuropathy (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 1 | 0
Petit mal epilepsy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 2
Radicular syndrome (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 4
Somnolence (Nervous system disorders) | 0 | 1
Spinal claudication (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 1
Syncope (Nervous system disorders) | 13 | 14
Syncope vasovagal (Nervous system disorders) | 1 | 3
Tension headache (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 12 | 14
Trigeminal neuralgia (Nervous system disorders) | 2 | 1
Vascular dementia (Nervous system disorders) | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 1 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 8 | 3
Anxiety (Psychiatric disorders) | 3 | 4
Confusional state (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 1 | 0
Delusional disorder, unspecified type (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 7 | 9
Depressive symptom (Psychiatric disorders) | 0 | 1
Dysthymic disorder (Psychiatric disorders) | 0 | 1
Hypochondriasis (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Stress (Psychiatric disorders) | 0 | 2
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 3 | 3
Calculus ureteric (Renal and urinary disorders) | 0 | 3
Haematuria (Renal and urinary disorders) | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 2
Nephritis (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 6 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 1
Renal cyst (Renal and urinary disorders) | 2 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 2
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 3
Urinary retention (Renal and urinary disorders) | 0 | 1
Adnexa uteri mass (Reproductive system and breast disorders) | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 1 | 0
Breast dysplasia (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 2
Cervical polyp (Reproductive system and breast disorders) | 1 | 2
Colpocele (Reproductive system and breast disorders) | 1 | 0
Cystocele (Reproductive system and breast disorders) | 4 | 5
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 1 | 1
Metrorrhagia (Reproductive system and breast disorders) | 2 | 1
Ovarian cyst (Reproductive system and breast disorders) | 6 | 2
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 3
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 3 | 4
Uterine prolapse (Reproductive system and breast disorders) | 8 | 8
Uterine synechiae (Reproductive system and breast disorders) | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 3 | 2
Vaginal fistula (Reproductive system and breast disorders) | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 15 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 14 | 11
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheobronchial dyskinesia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Scar (Skin and subcutaneous tissue disorders) | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 6
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Vasculitic rash (Skin and subcutaneous tissue disorders) | 1 | 0
Homicide (Social circumstances) | 0 | 1
Carpal tunnel decompression (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 5 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 3
Arterial haemorrhage (Vascular disorders) | 0 | 1
Arterial rupture (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 2 | 1
Arterial thrombosis (Vascular disorders) | 0 | 1
Arterial thrombosis limb (Vascular disorders) | 2 | 0
Arteriosclerosis (Vascular disorders) | 5 | 3
Arteriosclerosis obliterans (Vascular disorders) | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 5 | 9
Embolism (Vascular disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 0 | 2
Femoral artery occlusion (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 4 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 22 | 19
Hypertensive crisis (Vascular disorders) | 6 | 3
Hypotension (Vascular disorders) | 5 | 3
Hypovolaemic shock (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 2 | 1
Ischaemia (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 2
Peripheral embolism (Vascular disorders) | 0 | 2
Peripheral ischaemia (Vascular disorders) | 0 | 3
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 2
Superior vena caval occlusion (Vascular disorders) | 1 | 0
Temporal arteritis (Vascular disorders) | 2 | 0
Thrombophlebitis (Vascular disorders) | 1 | 3
Varicose vein (Vascular disorders) | 3 | 4
Vascular insufficiency (Vascular disorders) | 0 | 1
Vascular pseudoaneurysm (Vascular disorders) | 2 | 0
Vasculitis (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous stasis (Vascular disorders) | 1 | 1
Venous thrombosis limb (Vascular disorders) | 2 | 0
Wound haemorrhage (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3876) | Denosumab 60 mg Q6M (N=3886)
Cataract (Eye disorders) | 230 | 216
Constipation (Gastrointestinal disorders) | 356 | 351
Diarrhoea (Gastrointestinal disorders) | 231 | 224
Dyspepsia (Gastrointestinal disorders) | 209 | 175
Bronchitis (Infections and infestations) | 298 | 297
Cystitis (Infections and infestations) | 224 | 225
Influenza (Infections and infestations) | 334 | 331
Nasopharyngitis (Infections and infestations) | 600 | 563
Urinary tract infection (Infections and infestations) | 246 | 233
Fall (Injury, poisoning and procedural complications) | 233 | 190
Hypercholesterolaemia (Metabolism and nutrition disorders) | 236 | 280
Arthralgia (Musculoskeletal and connective tissue disorders) | 778 | 778
Back pain (Musculoskeletal and connective tissue disorders) | 1329 | 1340
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 289 | 295
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 397 | 383
Pain in extremity (Musculoskeletal and connective tissue disorders) | 430 | 450
Dizziness (Nervous system disorders) | 212 | 213
Headache (Nervous system disorders) | 255 | 234
Depression (Psychiatric disorders) | 217 | 206
Cough (Respiratory, thoracic and mediastinal disorders) | 238 | 224
Hypertension (Vascular disorders) | 619 | 603

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.